CLINICAL TRIAL: NCT05616039
Title: A Feasibility Randomised Controlled Study to Test the Use of Indocyanine Green Fluorescence Image-Guidance in Liver Surgery Compared to Standard Liver Surgery Alone in Reducing Microscopic Positive Tumour Resection Rate
Brief Title: I-FIGS Feasibility Study
Acronym: I-FIGS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Plymouth NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 317378
Record Dates: First submitted 2022-09-27; First posted 2022-11-14 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Liver Cancer; Hepatocellular Carcinoma; Liver Metastasis Colon Cancer
Keywords: Indocyanine green; Fluorescence Image Guided Surgery
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: Feasibility Randomized Controlled Study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Standard liver surgery) (Active Comparator): In this group, tumour/s, resection margin identification, and the type and number of liver resections will be based on naked eye examination, palpation, and intraoperative ultrasound. All the intra-operative findings will be recorded on a pre-designed proforma, and these details include the type of surgical approach (open, laparoscopic, and hand-assisted), if it is an open operation the type of incision, the location, number and size of tumour/s, relationship of the tumour/s to inflow and outflow of the liver, duration of surgery, and estimated blood loss. Post-operatively histology of the resected specimen including resection margin status will be recorded.
  Interventions: Procedure: Standard Liver Surgery
- Intervention Group (I-FIGS) (Experimental): Patients will receive intravenous indocyanine green(ICG) injection (0.03-0.05mg/kg) 2-4 hours before surgery. ICG comes in crystal form in 25mg dose. It will be diluted with 25ml of water, and the required dose as per the weight of the patient will be prepared freshly and given at least 2-4 hours before surgery. The surgical planning will be carried out as per the standard approach using the naked eye and IOUS. As for standard surgery, all intra-operative findings will be recorded on the proforma that contains the details that need to be collected. Once this is all recorded, ICG cameras will be switched on, and the additional findings (additional lesions detected, additional resections carried out) and change to surgical plan (change to the line of parenchymal transection) will be noted. Post-operatively histology of the resected specimen including resection margin status will be recorded.
  Interventions: Procedure: Standard Liver Surgery; Diagnostic Test: Indocyanine Fluorescent Image Guided Surgery (I-FIGS)

INTERVENTIONS:
Procedure: Standard Liver Surgery — Standard liver surgery using naked eye examination +/- palpation and intra-operative ultrasound scan (IOUS) examination to identify and remove liver tumours
Diagnostic Test: Indocyanine Fluorescent Image Guided Surgery (I-FIGS) — Use of I-FIGS in accurate identification of tumours and their margins
  Arms: Intervention Group (I-FIGS)

SUMMARY:
Background:

Removal of part of the liver (resection) is performed as a treatment for some cancers in the liver. To achieve the best possible outcomes, it is important that the cancer is removed completely (R0 resection) (1). Up to 30-50% patients develop recurrence within 2 years of surgery which could be due to incomplete removal of the cancer (2). Various techniques are used by the surgeons to identify the cancer tissue from the normal liver during the surgery so that it can be removed completely. These include examining with the naked eye, having a feel of the tumour, and performing an ultrasound scan. Even with these techniques it is difficult to identify the exact extent of the cancer. Also, the interpretation of the ultrasound scan can be subjective (3). A robust, objective, real-time navigation technique is required which can differentiate cancer from normal tissue.

Indocyanine green (ICG) is a dye which when given through the veins, is taken up and retained by cancer cells in the liver and they appear as fluorescent areas as compared to normal liver which appears dark. This principle can be used to identify the cancerous tissue accurately during the surgery and remove it completely (Indocyanine green Fluorescence Image-Guided Surgery: I-FIGS). It can also potentially detect additional tumours which were not identified before the surgery or during the surgery with standard techniques (4,5). However, there is a lack of good quality evidence on the usefulness of I-FIGS in liver surgery, so this needs to be tested in a large group of patients having liver surgery before any recommendations can be made.

Research Aim:

This initial study aims to assess whether a larger trial evaluating the role of I-FIGS in complete removal of the cancer tissue is feasible. Investigators will assess if patients are willing to take part in the study and whether they can gather relevant clinical outcome data from them all. Investigators will also gather patients' views about this novel technique and participating in the study.

Design and methods:

This study will involve 40 patients having planned liver surgery for liver tumour/s recruited from University Hospitals, Plymouth. Patients will be randomly allocated to have I-FIGS plus standard surgery or standard liver surgery alone. Patients in the I-FIGS group will have ICG injection 2-4 hrs prior to surgery (0.03-0.05mg/kg dose) on the day of surgery. The surgical planning will be carried out as per the standard approach using the naked eye and intra-operative ultrasound examination. Once this is all recorded, ICG cameras will be switched on, and the additional findings and change to surgical plan will be noted. Focus groups will explore participants experiences of being in the study. This will inform the design of the future larger trial.

Patient public involvement:

Investigators have involved patients who have had or are having liver surgery in the development of the study. Their views on the technique, trial procedures and outcome measures have been incorporated. They will continue to be involved and advise on the study.

Dissemination:

Results will be available via research journals and conferences.

ELIGIBILITY:
Inclusion Criteria:

• All adult patients (>16 years) requiring elective open/laparoscopic liver resection/s for liver metastases, primary hepatocellular and peripheral cholangiocarcinoma will be included in the study.

Exclusion Criteria:

* Patients allergic to iodine/contrast or shellfish
* Patients unable to consent to the study
* Patients with suspected liver adenomas and biliary cystadenomas
* Patients with suspected hilar cholangiocarcinoma
* Patients requiring emergency liver surgery
* Pregnant patients

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-11-23 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Feasibility outcomes | 10 weeks (from the day of recruitment till the histopathology report is available)
  * screening and recruitment rate
  * retention rate
  * adherence rates to study methods and procedures (consent, randomisation, intervention, data collection)
Clinical outcomes- Microscopic positive resection margin rate | From the day of surgery till the histopathology report is available (approximately 6 weeks)
  Number of patients with microscopic positive resection margins as compared to total number of patients, measured as percentage.
  Microscopic positive resection margin is defined as presence of tumour cells < 1 mm from the resection margin.

SECONDARY OUTCOMES:
Number of additional tumours detected | On the day of surgery
  Number of additional tumours detected by I-FIGS compared to Intra-operative ultrasound scan (IOUS) will be noted for each patient. A median value and range will be calculated for both the groups.
Duration of surgery | On the day of surgery
  This will be measured in minutes on the day of surgery. This will include the time from the time incision is taken (knife to skin) till the patient is extubated. A median value and range will be calculated for both the groups.
Post-operative length of stay | From the day of surgery till the day of discharge (approximately 10 days)
  This will be measured in number of days for each patient. A median value and range will be calculated for both the groups.
Complications | From the day of recruitment till the day of discharge (approximately 4 weeks)
  If case of any complications, these will be graded as per the Clavien-Dindo grading system.
  The unit of measure will be the Clavien-Dindo grade.

CONTACTS AND LOCATIONS:
Overall Officials: Somaiah Aroori, Study Director — University Hospitals Plymouth NHS Trust; Rahi Karmarkar, Principal Investigator — University Hospitals Plymouth NHS Trust
Locations (1):
- University Hospitals Plymouth NHS Trust, Plymouth, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No, we don not plan to share the raw individual patient data. However, the results of the study will be made available via research journals and conferences.

REFERENCES:
- [Background] Mise Y, Sakamoto Y, Ishizawa T, Kaneko J, Aoki T, Hasegawa K, Sugawara Y, Kokudo N. A worldwide survey of the current daily practice in liver surgery. Liver Cancer. 2013 Jan;2(1):55-66. doi: 10.1159/000346225. PMID 24159597
- [Background] Chan AWH, Zhong J, Berhane S, Toyoda H, Cucchetti A, Shi K, Tada T, Chong CCN, Xiang BD, Li LQ, Lai PBS, Mazzaferro V, Garcia-Finana M, Kudo M, Kumada T, Roayaie S, Johnson PJ. Development of pre and post-operative models to predict early recurrence of hepatocellular carcinoma after surgical resection. J Hepatol. 2018 Dec;69(6):1284-1293. doi: 10.1016/j.jhep.2018.08.027. Epub 2018 Sep 18. PMID 30236834
- [Background] Joo I. The role of intraoperative ultrasonography in the diagnosis and management of focal hepatic lesions. Ultrasonography. 2015 Oct;34(4):246-57. doi: 10.14366/usg.15014. Epub 2015 Apr 6. PMID 25971896
- [Background] Faybik P, Hetz H. Plasma disappearance rate of indocyanine green in liver dysfunction. Transplant Proc. 2006 Apr;38(3):801-2. doi: 10.1016/j.transproceed.2006.01.049. PMID 16647475
- [Background] Ishizawa T, Saiura A, Kokudo N. Clinical application of indocyanine green-fluorescence imaging during hepatectomy. Hepatobiliary Surg Nutr. 2016 Aug;5(4):322-8. doi: 10.21037/hbsn.2015.10.01. PMID 27500144